CLINICAL TRIAL: NCT06084286
Title: A Phase I, Open-label, Single-arm, Dose-escalation and Expansion Study of Specific Dual-targeting CLDN18.2 and PD-L1 CAR-T for Patients with CLDN18.2-positive Advanced Solid Tumors
Brief Title: Dual-targeting CLDN18.2 and PD-L1 CAR-T for Patients with CLDN18.2-positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director of Institute of Drug Clinical Trial of West China Hospital, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCART-007
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor
Keywords: CAR-T cell therapy; Solid Tumors; CLDN18.2-positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cell therapy (Experimental): Dual-targeting CLDN18.2 and PD-L1 CAR-T cells
  Interventions: Biological: Dual-targeting CLDN18.2 and PD-L1 CAR-T cells

INTERVENTIONS:
Biological: Dual-targeting CLDN18.2 and PD-L1 CAR-T cells — The trial consists of a traditional '3 + 3' pattern dose-escalation phase and a dose-expansion phase.

SUMMARY:
Claudin18.2(CLDN18.2) is a kind of integrin membrane protein in the tight junction between epithelium and endothelium, which is highly expressed in many solid tumors, especially in gastric cancer and pancreatic cancer. The CLDN18.2/PD-L1 dual-targeting CAR-T will be investigated in patients with CLDN18.2-positive advance solid tumors.

DETAILED DESCRIPTION:
In this study, the CLDN18.2/PD-L1 dual-targeting CAR-T cells will be injected intravenously to patients with CLDN18.2-positive advanced solid tumors, such as gastric adenocarcinoma or gastroesophageal junction adenocarcinoma and pancreatic adenocarcinoma, who had nearly no response to standard treatment. The safety and effectiveness will be evaluated. The safety evaluation standard refers to the standard of CTCAE 5.0. The evaluation standard of effectiveness refers to the evaluation standard of solid tumor curative effect RECIST 1.1 to evaluate the curative effect.

There are two phases of this study. The first is dose escalation phase, and 9 patients with CLDN18.2-positive advanced solid tumors are planned to be enrolled. The second is dose expansion phase. The curative effect has been observed in the first phase, and after the DLT observation period of the related dose group finished, the PI will decide whether to conduct the dose expansion research finally. It is planned to enroll 20 patients in dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age 18-75 years old;
2. Patients with pathologically/histologically confirmed diagnosis of solid tumors (such as advanced gastric adenocarcinoma or gastroesophageal junction adenocarcinoma and pancreatic adenocarcinoma) have received at least once systemic standard treatment and disease progressed; or refused/ cannot tolerate the subsequential standard treatment after the first line treatment;
3. Must have CLDN18.2-positive tumor expression ≥10% as determined by the CLDN18.2 IHC assay;
4. Estimated life expectancy > 3 months (according to investigator's judgement);
5. At least 1 measurable lesion per RECIST 1.1;
6. The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Sufficient venous access for leukapheresis collection and no other contraindications to leukapheresis;
8. Patients should have reasonable CBC counts, renal and hepatic functions;
9. No other serious diseases (autoimmune diseases or any immune deficiency disease);
10. Women of childbearing age must undergo a serum pregnancy test with negative results before screening and infusion and be willing to use effective and reliable method of contraception for at least 12-months after T-cell infusion;
11. Men must be willing to use effective and reliable method of contraception and are not allowed to donate sperm for at least 12-months after T-cell infusion;
12. Voluntarily participate in the research, understand and sign the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patient with hepatitis B or C active period, HIV infection ≥ the upper limit of the normal level;
3. Any uncontrolled active infection;
4. Patients who have clinically significant thyroid dysfunction;
5. Patients who have received prior cellular therapy such as CAR T, TCR, tumor-infiltrating lymphocytes;
6. Patients who are allergic to immunotherapy or any associated drugs, such as cytokines and the preconditioning regimen (cyclophosphamide, fludarabine);
7. Patients with untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression;
8. Patients have clinical significant cardiac conditions that researchers believe that participating in this clinical trial may endanger the health of the patients;
9. Unstable pulmonary embolism, deep venous embolism or other major arterial/venous thromboembolic events occurred within 6 months before enrollment;
10. Patients with active autoimmune diseases, history of autoimmune diseases or other diseases in need of immunosuppressive therapy;
11. Patients with major surgery or injury less than 4 weeks prior to leukapheresis or plan to have major surgery during the research period;
12. Patients with second malignancies in addition to targeted malignancies within 5 years before screening;
13. Patients with unstable/active ulcer or digestive tract bleeding;
14. Patient suffering from diseases that affect the signing of written informed consent or compliance with research procedures; or are unwilling or unable to comply with research requirements;
15. Patients who have a history or a tendency for digestive tract bleeding;
16. Patients who are inappropriate to participate in this research as considered by PI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 28 days
  Safety evaluation. AEs will be recorded and evaluated by CTCAE 5.0.
Dose-limiting toxicity (DLT) | 28 days
  Tolerability evaluation. DLT will be assessed by CTCAE 5.0.
Recommended phase II dose (RP2D) | Approximately 18 months
  Efficacy dose.

SECONDARY OUTCOMES:
Objective Remission Rate (ORR) | 3 months
  Include CR (complete response) and PR (partial response).
Progression-Free Survival (PFS) | Approximately 18 months
  The time from CAR-T administration to disease progression or death.
Duration of Control Rate (DCR) | Approximately 18 months
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Duration of Response (DOR) | Approximately 18 months
  It refers to the time from the first evaluation of CR or PR to the first evaluation of PD (Progressive Disease) or death from any reason.
Overall-Survival (OS) | Approximately 18 months
  It defined as the time from randomization to death from any cause, is a direct measure of clinical benefit to a patient. Patients alive or lost to follow-up are censored.
CAR-T cell numbers | 12 months
  Monitoring CAR-T cell numbers in blood to determine the persistence of CAR-T.
Anti-CAR antibody production | 12 months
  Immunogenicity
CAR-T cell phenotype | 12 months
  Immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: YongShen Wang, Prof., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheema PK, Burkes RL. Overall survival should be the primary endpoint in clinical trials for advanced non-small-cell lung cancer. Curr Oncol. 2013 Apr;20(2):e150-60. doi: 10.3747/co.20.1226. PMID 23559882
- [Background] Wagner DL, Fritsche E, Pulsipher MA, Ahmed N, Hamieh M, Hegde M, Ruella M, Savoldo B, Shah NN, Turtle CJ, Wayne AS, Abou-El-Enein M. Immunogenicity of CAR T cells in cancer therapy. Nat Rev Clin Oncol. 2021 Jun;18(6):379-393. doi: 10.1038/s41571-021-00476-2. Epub 2021 Feb 25. PMID 33633361